CLINICAL TRIAL: NCT02262195
Title: Dysfunctional Hemoglobin Pulse Co-ox
Brief Title: Dysfunctional Hemoglobin
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: QATP2338
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2014-10

CONDITIONS: Elevated Levels of Carboxyhemoglobin and Methemoglobin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Carboxyhemoglobin: Induced carboxyhemoglobin levels up tp 15 percent.
  Interventions: Other: Elevated levels of carboxyhemoglobin
- Methemoglobin: Induced methemoglobin levels up to 15 percent.
  Interventions: Other: Elevated levels of carboxyhemoglobin

INTERVENTIONS:
Other: Elevated levels of carboxyhemoglobin — Comparison of pulse co-oximeters
  Other Names: Elevated levels of methemoglobin

SUMMARY:
The purpose of the study is to determine if a new pulse oximeter accurately detects carboxyhemoglobin and methemoglobin when intentionally increased in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Subjects does not have significant medical problems
* Subject is willing to provide written informed consent
* Subject is between 18 and 45 years of age

Exclusion Criteria:

* Has a BMI greater than 31
* Has had any relevant injury at the sensor location site
* Has deformities or abnormalities that may prevent proper application of the device under test
* Has a known respiratory condition
* Is currently a smoker
* Has a known heart or cardiovascular condition
* Is currently pregnant
* Is female and actively trying to get pregnant
* Has a clotting disorder
* Is known to have a hemoglobinopathy such as (anemia, bilirubinemia, sickle-cell anemia, inherited or congenital methemoglobinemia)
* The subject has a COHb greater than 3% or MetHb greater than 2%
* Has taken blood thinners or medication with aspirin within the last 24 hours
* Has unacceptable collateral circulation from the ulnar artery
* Has donated more than 300 mL of blood within one month prior to start of study
* Is unwilling or unable to provide written informed consent to participate in the study
* Is unwilling or unable to comply with the study procedures
* Has another health condition which in the opinion of the principal investigator makes him/her unsuitable for testing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Evaluate carboxyhemoglobin over the range of 0-15 percent as assessed by co-oximetry | 4 hours
Evaluate methemoglobin over the range of 0-15 percent as assessed by co-oximetry | 4 hours

SECONDARY OUTCOMES:
Determine oxygen saturation accuracy in conditions of elevated carboxyhemoglobin | 4 hours
Determine oxygen saturation accuracy in conditions of elevated methemoglobin | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Phillip E Bickler, MD, PhD, Principal Investigator — University of San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States